CLINICAL TRIAL: NCT05901753
Title: A Comparative Study Between Laryseal Pro Supra Glottic Device (SGD) With Proseal Laryngeal Mask Airway Regarding Clinical Performance in Patients Undergoing Ophthalmic Surgery. A Prospective Randomized Control Study
Brief Title: A Comparative Study Between Laryseal Pro Supra Glottic Device (SGD) With Proseal Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MS-631-2022
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ophthalmic Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside.
  This study will be performed by 2 investigators; the first one (implementing doctor) who will insert supra glottic airway device based on patients' weight as per the manufacturers' size recommendations and according to a computer-generated sequence of random numbers and sealed envelope. The second anesthetists (planning doctor) will be blinded to the technique performed, and will monitor the patients intra and postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryseal pro supra glottic device (SGD) (Experimental): Laryseal pro SGD, the jaw will be lifted during insertion and the head will be extended, proper lubrication of both the front and back of the laryseal pro as if the patient's mouth is dry the laryseal pro ridges can get hung up on the back of the tongue during placement.
  Interventions: Device: Laryseal pro supra glottic device
- Laryngeal Mask Airway- Proseal™ (Experimental): The LMA-Proseal™ will be inserted using the digit method. The size will be determined according to the patient's weight and inserted according to the manufacture's recommendation with the use of an introducer.
  Interventions: Device: Laryngeal Mask Airway- Proseal™

INTERVENTIONS:
Device: Laryseal pro supra glottic device — The laryseal pro SP will be advanced at a forward angle aiming for the back of the tongue and soft palate. Then the colored connector will be pushed by index finger till feeling resistance . Device insertion will be considered successful by observing bilateral chest wall movement as well as a stable square-wave capnogram trace
  Other Names: supra glottic device
  Arms: Laryseal pro supra glottic device (SGD)
Device: Laryngeal Mask Airway- Proseal™ — The cuff will be inflated with air and the cuff's pressure will be adjusted to 70 mmHg using a cuff pressure manometer. the device will be lubricated well on both sides, head and neck were placed in neutral position, the proximal firmer part of the device will be compressed between the thumb and two fingers and advanced toward hard and soft palate, the tab will be pulled slightly if needed to increase curvature of the device for better fitting, the device will be advanced till resistance felt.
  Other Names: supra glottic device
  Arms: Laryngeal Mask Airway- Proseal™

SUMMARY:
Difficult airway is a nightmare to every anesthetist. Over the last decade, several supraglottic airway devices appeared in the clinical field as an alternative to the more invasive endotracheal intubation(1). However, many anesthetists found themselves unaccustomed with the newly invented devices .Supraglottic airway devices (SAD) have become valuable for both routine and difficult airway management. After the creation of the laryngeal mask airway (LMA) classic in the 1980s, there has been a steady increase in the applications for use of supraglottic airways. Developed by Dr. Archie Brain in 2000, the ProSeal laryngeal mask airway (P-LMA) is a second-generation supraglottic airway device (SAD) with two lumens separating the alimentary and respiratory channels from each other This study aim to compare the use of the Laryseal Pro and the Proseal LMA as a supraglottic devices by measuring the time of insertion (which is defined as time interval in seconds between removing the ventilation mask and picking the device up till connecting to the ventilator and appearance of the ﬁrst wave on the capnogram)

Objectives:

To determine ease of insertion for each supra glotic device. To Estimate the time needed for insertion for each supra glotic device. To identify airway pressure leakage, gastric tube insertion success and complication for each device.

It is hypothesized that the Laryseal pro is a safe superior supraglottic airway device and its insertion is easier than the LMA-Proseal .

DETAILED DESCRIPTION:
This a randomized control trial is designed to include (120) patients ASA physical status I ,II patients ranging from(18) to(60)years old scheduled for ophthalmic surgery

Patients meeting the inclusion criteria will be randomly assigned to receive either:

Group A: Laryseal pro supra glottic device (SGD) (n=60) Group B: Laryngeal Mask Airway- Proseal™ (n=60) Anesthesia management

Preoperative procedures:

After being accepted into the study, participants age, gender, weight, medications and any other co morbidities will be collected. patients will be allowed to fast for 6-8 h before surgery.

After securing IV access by 20G cannula, all patients will receive 0.05mg/kg midazolam for anxiety. Ranitidine 50mg, metoclopramide 10mg and intravenous atropine 0.01 mg/kg as a premedication. Routine monitoring devices will be installed (basline blood pressure, heart rate, and pulse oximetry data) Proper airway assessment of the patients will be done according to El-Ganzouri Airway Scoring System(13) Intraoperative monitoring includes ASA standard monitoring Electrocardiography (ECG), noninvasive blood pressure, pulse oximetry for O2 saturation, end-tidal CO2 values by capnography

Intraoperative procedures:

Induction of general anaesthesia will be achieved by approximate doses according to ideal body weight of Fentanyl 1ug/kg, Propofol 2mg/kg and Atracurium 0.5mg/kg and Lidocaine 1mg/kg , 3 minutes of for oxygenation and mask ventilation before device insertion .

Anesthesia maintenance will be achieved with the randomly assigned supraglottic device for each group which will be inserted and reconnected to the ventilator circuit., 2 minumium alveolar concentration of sevoflurane, volume-controlled mode ventilation, respiratory rate will be adjusted according to Et CO2 to range between 35-40 mmHg, a tidal volume of 6-8 ml/kg and mixture of gases in proportion 50% oxygen and 50% air

The LMA-Proseal™ will be inserted using the digit method. The size will be determined according to the patient's weight and inserted according to the manufacture's recommendation (12) with the use of an introducer. The cuff will be inflated with air and the cuff's pressure will be adjusted to 70 mmHg using a cuff pressure manometer. the device will be lubricated well on both sides, head and neck were placed in neutral position, the proximal firmer part of the device will be compressed between the thumb and two fingers and advanced toward hard and soft palate, the tab will be pulled slightly if needed to increase curvature of the device for better fitting, the device will be advanced till resistance felt.

For Laryseal pro SGD, the jaw will be lifted during insertion and the head will be extended, proper lubrication of both the front and back of the laryseal pro as if the patient's mouth is dry the laryseal pro ridges can get hung up on the back of the tongue during placement. The laryseal pro SP will be advanced at a forward angle aiming for the back of the tongue and soft palate. Then the colored connector will be pushed by index finger till feeling resistance . Device insertion will be considered successful by observing bilateral chest wall movement as well as a stable square-wave capnogram trace. Failed device placement will be defined as being unable to observe a smooth square-wave capnograph, inadequate ventilation, no rise of the chest wall, and significant leakage from the gastric drain tube If, after two attempts, the device not properly inserted, endotracheal intubation will be done and those patients will be excluded from the study.

Insertion time of the study device will be recorded for each device which is defined as time interval between picking the device up till appearance of the ﬁrst wave on the capnogram.

The ease of insertion will be classified based on insertion attempts (1 = first attempt, 2 = second attempt, 3 = third attempt, 4 = impossible) The vital signs(heart rate and mean blood pressure) will be recorded; just prior to device insertion (T1); after connection to capnography (T2), to assess the pressor response during device insertion The airway seal pressure will be assessed for each device , measured with head in the neutral position, under manual ventilation by closing the adjustable pressure-limiting (APL) valve to 30 cmH2O adjustable pressure-limiting (APL) valve to 30 cmH2O at a fixed gas flow of 3 L.min-1 , 7, and observing of the rise of the ventilator's airway pressure[14]. A "puffing" sound will be heard near the patient's mouth (release of pressure) indicating the airway seal pressure.

Once patients reconnected to the ventilator circuit, a gastric tube will be introduced through the integrated drainage channel present in both devices. To standardize the technique, the same brand gastric tube will be used for both devices. The success rate of its insertion will be recorded. Ease of gastric tube insertion will be graded on a three-point scale (1 = first attempt, 2 = second attempt and 3 = impossible). After venting the stomach the blocker will be introduced and inflated to achieve proper sealing. The surgery will be allowed to proceed after ensuring proper positioning and sealing of the device.

At the end of surgery, adequate reversal of residual neuromuscular blockade will be achieved The device will be removed and checked for any blood streaked mucous as a sign of airway trauma. Post-operative sore throat or hoarseness of voice will be assessed at 0, 2 and 4 h. Any regurgitation , pulmonary aspiration, bronchospasm , hypoxemia will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* Age 18-60 years
* GANZOURI airway scores less than 4
* Patients undergoing ophthalmic surgeries not exceeding two hours under general anesthesia (cataract surgery,glaucoma surgery, corneal transplant, strabismus surgery

Exclusion Criteria:

* Patients have risks of gastric aspiration (patients known to have gastro esophageal reflux disease (GERD), hiatus hernia or previous upper gastrointestinal tract surgery)
* patients have respiratory or pharyngeal pathology
* morbidly obese patients with body mass index >40 kg/m3

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
The time of insertion of supra glottic device | time interval between picking the device up till appearance of the ﬁrst wave on the capnogram. (seconds)
  time interval between picking the device up till appearance of the ﬁrst wave on the capnogram

SECONDARY OUTCOMES:
complications | it will be measured postoperatively at 0, 3, 6 hours
  Blood on device after removal, vomiting, aspiration, bronchospasm and Post-operative sore throat or hoarseness of voice

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ismael, professor, Study Director — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No